CLINICAL TRIAL: NCT04213534
Title: The Influence of Urate-lowering Therapy on Sperm Quality of Male Gouty Patients：A Prospective Cohort Study
Acronym: INITIAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Jinxia Zhao, Deputy department director, Peking University Third Hospital
Other Study IDs: M2019259
Record Dates: First submitted 2019-12-20; First posted 2019-12-30 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Gout
Keywords: gout; management; semen quality; male fertility; allopurinol; febuxostat; benzbromarone
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gout is a kind of crystal-associated arthropathy caused by monosodium urate deposition, which is directly related to hyperuricemia caused by purine metabolic disorder and/or decreased uric acid excretion. It belongs to the category of metabolic rheumatism. Gout can be complicated with kidney disease. The severe cases can occur joint destruction, renal function damage, and often accompanied by hyperlipidemia, hypertension, diabetes, arteriosclerosis and coronary heart disease and so on.

The prevalence of gout varies greatly from different countries. But on the whole, the prevalence of gout is increasing year by year, and the incidence of gout is getting younger. With the continuous improvement of living standards in today's society, middle-aged men have quietly become a high incidence group of gout.

The pathophysiological basis of gout is hyperuricemia, so reducing uric acid is the core of gout treatment. The reducing uric acid in patients with gout is a long-term process, and the drug can not be stopped after the serum uric acid is reduced to normal. Once patients with gout stop taking uric acid-lowering drugs, serum uric acid quickly returns to the pre-treatment level, which can not only cause gout attack again, but also bring the risk of kidney and cardio-cerebrovascular involvement if serum uric acid does not reach the control standard for a long time. Therefore, uric acid-lowering therapy requires the use of a minimum dose of uric acid-lowering drugs to maintain long-term uric acid levels.

In recent years, with the aggravation of environmental pollution and the postponement of childbearing age, the incidence of male infertility is increasing year by year. However, there are relatively few studies on the effect of gout caused by hyperuricemia on male sperm quality. With the rejuvenation of gout patients and the long-term nature of uric acid-lowering therapy, the safety of uric acid-lowering drugs in male gout patients of childbearing age during pregnancy is not sure. Coupled with the opening of China's comprehensive second-child policy, more and more male gout patients join this fertility group. Unfortunately, so far, no animal or human trial has observed the effect of uric acid-lowering drugs on sperm quality. For this reason, this study intends to carry out this observational clinical trial to evaluate the effect of long-term use of uric acid-lowering drugs on male sperm quality by collecting relevant data of patients with gout treated with uric acid-lowering drugs. Aim to provide a theoretical basis for the safety of uric acid-lowering drugs during pregnancy.

DETAILED DESCRIPTION:
1. Research drugs. Three kinds of uric acid lowering drugs, allopurinol, febuxostat and benzbromarone, will be evaluated in this study.
2. Study design and sample size calculation. This study was designed as a single-center prospective cohort study. After a careful search of the relevant literature, there are no reports of similar studies, so it is impossible to accurately estimate the sample size. Therefore, this study planned to enroll 20 patients with gout who were using allopurinol, febuxostat and benzbromarone to reduce uric acid, respectively. It is planned to recruit 5 gouty patients and 5 control males every month. Therefore, the whole study needs to last at least 12 months after initiation
3. Research process. The process of this study does not affect the routine diagnosis and treatment procedures of patients with gout. Our research team is made up of doctors majoring in rheumatology and andrology. Therefore, we can make routine clinical diagnosis and treatment according to the specific conditions of patients with gout.

1) Screening period. It will takes about 2 weeks, including the following forms:

1. Patients with gout are in acute attack. According to the guidelines for the diagnosis and treatment of gout, we should first give them anti-inflammatory and analgesic treatment. Non-steroidal anti-inflammatory drugs(NSAIDs) or colchicine can be selected to control acute symptoms. Then we performed the semen analysis after the joint swelling and pain is completely improved. If the patient meets our admission criteria, urate-lowering therapy should be initiated according to the clinical practice. And we regard this time as week 0. NSAIDs or colchicine can be prophylacticly used for at least 2 weeks combined with urate-lowering treatment in case of gout flare.
2. Patients with gout in remission. For this kind of patients, we directly conduct semen analysis. If the results meets our admission criteria, urate-lowering therapy should be initiated according to the clinical practice. We also regard this time as week 0. And the preventive use of NSAIDs or colchicine is the same as above.

   2) Follow-up stage. The follow-up cycle was calculated after the beginning of urate-lowering therapy. We will detect the blood routine, urine routine, liver and kidney function and serum uric acid at the time of screening and week 2, week 4, week 8 and week 12 visits. The patients will receive the repeated sperm analysis at week 4 and week 12, respectively. At the same time, we will collect all the corresponding data on the case report form.

   4、Patient withdrawal. Patients can drop out of the trial at any time. Researchers can also persuade patients to withdraw for a variety of reasons, including baseline screening for sperm quality below World Health Organization (WHO) standards, adverse events, safety concerns, or patients' failure to comply with the trial regimen.

   5、Eliminated cases. For some reason, those who are not completed as planned and whose observation records are incomplete are eliminated cases. Those who are interrupted due to serious adverse reactions should be regarded as cases of adverse reactions and shall not be included in the statistics of comparative analysis of semen.

   6、Treatment regimen. Baseline screening: if the patient meets the selection criteria and is not in the gout attack period, we can consider the direct start of uric acid-lowering drug treatment. The choice of uric acid-lowering drugs should be based on the patient's drug use taboos for real-world choice. If the patient is in the attack stage of acute arthritis, we need to control the acute symptoms, and we can consider using NSAIDs, and then start the uric acid treatment after the joint symptoms are completely improved.

Uric acid-lowering therapy: the beginning of uric acid-lowering therapy must be combined with NSAIDs or colchicine to prevent gout.

* Allopurinol, the initial dose of 125mg once a day. If serum uric acid is not less than 360 µm/L after 4 weeks, the dose can be increased to 250mg once a day, and the highest dose does not exceed 500mg every day.

  * Febuxostat, the initial dose of 20mg once a day. If serum uric acid is not less than 360 µm/L after 4 weeks, the dose can be increased to 40mg once a day, and the highest dose does not exceed 80mg every day.

    * Benzbromarone, the initial dose of 25mg once a day. If serum uric acid is not less than 360 µm/L after 4 weeks, the dose can be increased to 50mg once a day, and the highest dose does not exceed 100mg every day.

      7、Assessment. We will use two methods to assess male fertility: basic semen analysis and sperm DNA integrity analysis.
      1. Basic semen analysis and sperm DNA fragmentation were performed at Reproductive Medicine Centre, Peking University Third Hospital using standard laboratory procedures, per WHO guidelines (2010 5th edition). This is a microscopic evaluation of fresh semen that assesses sperm concentration, viability, motility, and morphology.
      2. Sperm Testing for DNA Fragmentation:

         The sperm DNA fragmentation assay was utilized to assess sperm DNA integrity based upon the literature report (Cytometry 1985; 6(3): 238-53) in which sperm DNA is stained with acridine orange and analyzed by flow cytometry.Two measurements are then produced: %DFI (DNA fragmentation index) which indicates level of sperm DNA breaks and %HDS (high DNA stainability) which is reported to correlate to levels of immature sperm and somatic cells such as white blood cells.
      3. Serum samples for the analysis of serum uric acid were collected at the time of screening, week 4, week 8 and week 12, or early termination.

         8、Samples collection, preservation and destruction

      a. Semen samples were collected by masturbation after an instructed period of 2 to 3 days without ejaculation in the semen collection room of Peking University third Hospital after signing the informed consent according to the trial scheme. After semen liquefaction (30 minutes to 1 hour), an aliquot was used for semen analysis and a second aliquot of raw semen was frozen within 2 hours of collection at -80° C.

      b. Semen samples are uniformly preserved until destroyed after the end of this trial. The test time is expected to be 2-3 years.

      c. At the end of the trial, the semen samples were uniformly destroyed. The frozen semen was reheated at room temperature and completely soaked in 0.5% sodium hypochlorite disinfectant. Finally, the disinfection solution containing semen was treated as medical waste.

      9、Quality control.

      a. Carry out publicity and education to the subjects to reduce the rate of loss of follow-up; b. Semen quality analysis system was used to detect semen quality indexes such as sperm density, motility, forward motility ratio and so on. Quality control of standard samples was carried out for every 10 samples tested.

      10、Statistical analysis. We will use SPSS 20.0 software for statistical analysis. All statistical tests are bilateral test, P value less than or equal to 0.05 will be considered to be statistically significant. When comparing the difference of curative effect between the parameters before and after gout treatment, paired t-test was used if the measurement data were in accordance with normal distribution. Independent sample t-test was used for comparison among different intervention groups. Nonparametric test is used if the measurement data do not conform to the normal distribution. Chi-square test was used to compare the counting data between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male, aged 18 ~45 years old;
2. In accordance with the gout classification criteria of the American Rheumatic Society in 1977 or ACR/EULAR (European Alliance against Rheumatism) in 2015 ;
3. Willing to receive uric acid-lowering drugs regularly for at least 3 months;
4. No drugs affecting sperm quality were taken within 3 months before screening.
5. Sign the informed consent form.

Exclusion Criteria:

1. Patients who have a pregnancy plan during the trial;
2. Patients with severe heart, liver, kidney and other important organs, blood and endocrine system diseases, the evaluation criteria are as follows:

   1. Heart disease: patients with a history of heart disease such as decompensated cardiac insufficiency, refractory hypertension or coronary heart disease;
   2. Liver function: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal reference value (ULN);
   3. Renal function: complicated with renal tubule and/or renal interstitial lesions, or renal insufficiency: serum creatinine≥ULN or glomerular filtration rate (eGFR) <60ml/min/1.73m2;
3. leukocyte (WBC) count <3 × 109/L and/or hemoglobin (Hb) <100g/L and/or platelet (PLT) count <80 × 109/L;
4. Other serious diseases, such as tumors, etc;
5. Those who are unable to cooperate with the treatment of mental illness or other reasons;
6. Allergic constitution or multi-drug allergy;
7. Those who are known to be allergic or intolerant to uric acid-lowering drugs in the trial;
8. Chromosome abnormality or deletion of AZF region of Y chromosome;
9. Previous history of orchitis, epididymitis, mumps or varicocele affecting sperm quality;
10. Positive semen bacterial culture, or Chlamydia trachomatis, Ureaplasma Urealyticum and Mycoplasma hominis;
11. Those who have a history of exposure to high temperature, chemistry, physics or toxicants in the past year;
12. Those who undergo X-ray or CT examination in the past 3 months and during the period of enrollment;
13. Patients with other systemic diseases who are being treated with other drugs that may affect semen quality.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The purpose of this study is to investigate the effect of uric acid-lowering drugs on sperm quality, so the inclusion of patients must be male.
Study Population: The patients included in this study are male patients with gout. These patients were treated in the outpatient clinic of the Department of Rheumatology and Immunology, Peking University Third Hospital, China. And they were followed up regularly in the outpatient clinic. We will give individualized uric acid lowering treatment according to the specific conditions of the patients on the basis of clinical routine. Then the effect of uric acid-lowering drugs on semen quality parameters was observed.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The mean change from baseline to week 12 in semen quality. | At baseline, week 4 and week 12 visits
  According to the current world health orgnization semen analysis guidelines, semen quality evaluation can not use a single index to evaluate semen quality grade. The change of semen quality needs to be evaluated comprehensively from two aspects, namely basic semen analysis and sperm DNA integrity analysis Therefore, all the measurements will be aggregated to arrive at the reported value as semen quality.

SECONDARY OUTCOMES:
Comparison of the reproductive hormone levels, oxidative stress level,the rate of the target serum urate level of <6.0 mg/dl at week12 of treatment, et al among different groups. | At baseline, week 4 and week 12 visits

CONTACTS AND LOCATIONS:
Overall Officials: Jinxia Zhao, doctorate, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China